CLINICAL TRIAL: NCT06188130
Title: The Effect of rTMS and tDCS Treatments Combined With Robotic Rehabilitation on Gait and Motor Recovery in Partial Chronic Spinal Cord Injury
Brief Title: The Effects of rTMS and tDCS Combined With Robotic Rehabilitation In Patients With Spinal Cord Injury
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Ankara City Hospital Bilkent (Other)
Responsible Party: Principal Investigator, Emre Adıgüzel, Emre Adıgüzel, Associate professor, Ankara City Hospital Bilkent, Ankara City Hospital Bilkent
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10025144
Record Dates: First submitted 2023-08-24; First posted 2024-01-03 (Actual); Last update posted 2024-01-03 (Actual); Status verified 2023-08

CONDITIONS: Chronic Spinal Cord Disorder

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- active rTMS (Experimental): Participants recevied 20 Hz high frequency repetetive TMS during 20 minutes and a total of 1200 stimuli for 15 sessions. The patient received robotic therapy for lower extremity just after each active TMS sessions
  Interventions: Other: active rTMS
- sham rTMS (Sham Comparator): Participants recevied sham TMS during 20 minutes and a total of 1200 sham stimuli for 15 sessions with sham coil. The patient received robotic therapy for lower extremity just after each sham TMS sessions
  Interventions: Other: sham rTMS
- active tDCS (Experimental): Participants recevied 2 mA anodal transcranial direct current stimulation 20 minutes for 15 sessions. The patient received robotic therapy for lower extremity just after each active tDCS sessions
  Interventions: Other: active tDCS
- sham tDCS (Sham Comparator): Participants recevied sham stimulation. The patient received robotic therapy for upper extremity just after each sham tDCS sessions
  Interventions: Other: sham tDCS

INTERVENTIONS:
Other: active rTMS — Participants recevied 20 Hz high frequency repetetive TMS during 20 minutes and a total of 1200 stimuli for 15 sessions. Motor threshold was defined as the minimum stimulus intensity eliciting 5 responses of about 50 µV out of 10 consecutive trials (50% successful MEPS) in the relaxed dominant side abductor pollicis brevis (APB).The patient received robotic therapy for lower extremity just after each active TMS sessions.
  Arms: active rTMS
Other: sham rTMS — Participants recevied sham TMS during 20 minutes and a total of 1200 sham stimuli for 15 sessions with sham coil employed was identical in shape and size to the real stimulation coil and produced no magnetic field. The patient received robotic therapy for lower extremity just after each sham TMS sessions.
  Arms: sham rTMS
Other: active tDCS — Participants recevied 2 mA anodal transcranial direct current stimulation 20 minutes for 15 sessions.The electrodes will be placed anodal to the Cz central (International 10/20 Electroencephalogram System) area, corresponding to the location of the dominant hemisphere lower extremity motor cortex and cathodal to the contralateral supraorbital region. The patient received robotic therapy for lower extremity just after each active tDCS sessions.
  Arms: active tDCS
Other: sham tDCS — Participants recevied sham stimulation were applied current was ramped up either over 10 seconds, with an equal amount of time for tapering off. The patient received robotic therapy for lower extremity just after each sham tDCS sessions
  Arms: sham tDCS

SUMMARY:
The purpose of this study is to assess the effect of rTMS and tDCS combined with robotic therapy on motor functional recovery and gait parameters

DETAILED DESCRIPTION:
After being informed about study and potential risks, all patient giving written informed consent will undergo screening period determine eligibility for study entry. The patients who meet the eligibility requirements will be randomized into four groups in a 1:1 ratio to active rTMS, sham rTMS, active tDCS and sham tDCS.

ELIGIBILITY:
Inclusion Criteria:

* Having traumatic SCI
* Between 6 months and 2 years after SCI
* 18-65 years old
* Signing an informed consent form showing his/her consent to participate in the study.
* Motor incomplete cervical or thoracic SCI
* Spasticity in the lower extremity ≤2 according to the Modified Ashworth Scale

Exclusion Criteria:

* History of epilepsy
* A cardiac pacemaker
* Pregnancy
* Neurological diseases other than SCI
* Metallic implant in brain or scalp (including cochlear implant)
* Previous brain surgery
* Orthopedic disease that prevents lower extremity movements
* Diagnosis of malignancy
* Receiving robotic /TMS/tDCS treatments in the last 6 months

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2023-12-30 (Estimated); Study Completion 2024-01-15 (Estimated)

PRIMARY OUTCOMES:
Lower extremity motor scores according to ASIA examination | initial, 3th week 9th week changes
  ASIA (American Spinal Injury Association) Classification System is used to assess and determine the neurological status of individuals with spinal cord injuries. This classification system consists of five different classes:
  ASIA A:There is complete loss of motor and sensory function. ASIA B:Sensation is present in the sacral region (S4-S5), but motor function loss persists.
  ASIA C:Motor function loss persists, but there is observable muscle contraction (muscle strength) in specific muscle groups.
  ASIA D:Motor function loss continues, but uncontrolled movements can be observed.
  ASIA E:Normal sensory and motor functions are present.
  The ASIA classification is a widely used system for evaluating the severity and effects of spinal cord injuries. This classification provides important guidance for the planning of treatment and rehabilitation processes.
Walking Index for SCI - II (WISCI-II) | initial, 3th week 9th week changes
  Physical limitation for walking secondary to impairment is defined at the person level and indicates the ability of a person to walk after spinal cord injury. The development of this assessment index required a rank ordering along a dimension of impairment, from the level of most severe impairment (0) to least severe impairment (20) based on the use of devices, braces and physical assistance of one or more persons. The order of the levels suggests each successive level is a less impaired level than the former. The ranking of severity is based on the severity of the impairment and not on functional independence in the environment.
10 meter walking test | initial, 3th week 9th week changes
  The 10 Metre Walk Test is a performance measure used to assess walking speed in meters per second over a short distance[1]. It can be employed to determine functional mobility and gait.

SECONDARY OUTCOMES:
Modified Ashworth Scale | initial, 3th week 9th week changes
  İts performed by extending the patients limb first from a position of maximal possible flexion to maximal possible extension ( the point at which the first soft resistance is met). Afterwards, the modified Ashworth scale is assessed while moving from extension to flexion
  0 No increase in tone
  1 slight increase in tone giving a catch when slight increase in muscle tone, manifested by the limb was moved in flexion or extension.
  1+ slight increase in muscle tone, manifested by a catch followed by minimal resistance throughout (ROM ) 2 more marked increase in tone but more marked increased in muscle tone through most limb easily flexed 3 considerable increase in tone, passive movement difficult 4 limb rigid in flexion or extension
Visual Analogue Scale | initial, 3th week 9th week changes
  The Visual Analogue Scale (VAS) measures pain intensity. The VAS consists of a 10cm line, with two end points representing 0 (no pain) and 10 (pain as bad as it could possibly be).

CONTACTS AND LOCATIONS:
Overall Officials: Emre Adıgüzel, Principal Investigator — Ankara City Hospital Bilkent
Locations (1):
- Ankara Bilkent City Hospital Pyhsical Treatment and Rehabilitation Hospital, Ankara, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No